CLINICAL TRIAL: NCT03547206
Title: A Double-Masked Clinical Study Evaluating the Efficacy and Safety of RPh201 Treatment in Participants With Previous NAION
Brief Title: Efficacy & Safety of RPh201 Treatment in Patients With Previous Nonarteritic Anterior Ischemic Optic Neuropathy (NAION)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated by Sponsor
Sponsor: Regenera Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RGN-ON-002
Record Dates: First submitted 2018-05-24; First posted 2018-06-06 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Nonarteritic Anterior Ischemic Optic Neuropathy
Keywords: NAION; ischemic optic neuropathy
MeSH Terms: conditions — Optic Neuropathy, Ischemic | interventions — Cottonseed Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All clinic staff and participants will be masked to group assignments. Only the Data and Safety Monitoring Board (DSMB) and designated unmasked staff at the Coordinating Center will have access to the group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- RPh201 Cohort A (Experimental): A 26-week schedule consisting of twice-weekly subcutaneous administration of 400 μL of the Investigational Medical Product (IMP) (20 mg RPh201).
  Interventions: Drug: RPh201 Cohort A
- Placebo Cohort A (Placebo Comparator): A 26-week schedule consisting of twice-weekly subcutaneous administration of 400 μL of the vehicle control.
  Interventions: Other: Placebo Cohort A
- RPh201 Cohort B (Experimental): A 12-week schedule consisting of four-times-per-week subcutaneous administration of 400 μL of the Investigational Medical Product (IMP) (20 mg RPh201).
  Interventions: Drug: RPh201 Cohort B
- Placebo Cohort B (Placebo Comparator): A 12-week schedule consisting of four-times-per-week subcutaneous administration of 400 μL of the vehicle control.
  Interventions: Other: Placebo Cohort B

INTERVENTIONS:
Drug: RPh201 Cohort A — RPh201 is a proprietary, isolated botanical extract of gum mastic for treatment of nonarteritic anterior ischemic optic neuropathy (NAION).
  Arms: RPh201 Cohort A
Other: Placebo Cohort A — The placebo is composed of RPh-201 excipients (cottonseed oil stabilized with butylated hydroxytoluene [BHT]).
  Other Names: Cottonseed oil
  Arms: Placebo Cohort A
Drug: RPh201 Cohort B — RPh201 is a proprietary, isolated botanical extract of gum mastic for treatment of nonarteritic anterior ischemic optic neuropathy (NAION).
  Arms: RPh201 Cohort B
Other: Placebo Cohort B — The placebo is composed of RPh-201 excipients (cottonseed oil stabilized with butylated hydroxytoluene [BHT]).
  Arms: Placebo Cohort B

SUMMARY:
This study is designed as a double-masked, randomized, placebo-controlled, clinical study to evaluate the efficacy and safety of subcutaneous (SC) administration of RPh201 in participants with previous NAION. All participants enrolled in Cohort A of the study will have a documented history of NAION for at least 12 months and at most, five years prior to enrollment. Participants enrolled in Cohort B of the study will have a documented history of NAION for at least 6 months and at most, three years prior to enrollment.

DETAILED DESCRIPTION:
This study is designed as a double-masked, randomized, placebo-controlled, clinical study to evaluate the efficacy and safety of SC administration of RPh201 in participants with previous NAION.

Following a screening phase of 1-8 weeks, participants will attend a baseline visit in which they will undergo testing and visual function assessments. Participants then will be randomized to receive RPh201 or control.

Cohort A After randomization, participants will begin a 26-week schedule consisting of twice-weekly treatment. Participants will return to the clinic for visits at Week 1, Week 4, Week 12 and Week 26 and Week 52

Cohort B After randomization, participants will begin a 12-week schedule consisting of four-times-per-week treatment. Participants will return to the clinic for visits at Week 4 and Week 12.

Safety and efficacy parameters will be recorded throughout the duration of the study.

ELIGIBILITY:
Inclusion Criteria (Cohort A):

1. The participant must be 50 years of age or older at the time of the NAION episode in the study eye. This means that the participant's age at enrollment must be greater than or equal to the sum of 50 plus the number of years since NAION (e.g., at least 52 years of age if the episode was two years prior).
2. The participant must understand the nature of the procedure and provide written informed consent prior to any study procedure.
3. The participant has a definitive clinical diagnosis of NAION in the study eye that developed at least 12 months before randomization. Specifically, the disc swelling must have been observed and documented (by examination, OCT or photograph) by an ophthalmologist or neuro-ophthalmologist who previously examined the participant at the time of the NAION episode in the study eye during the acute episode.
4. The participant's study eye must have disc pallor (global or segmental) present.
5. The participant's study eye must have stable visual acuity (see Sections 5.3.3 and 5.3.4).
6. Using the study eye, the participant must read at least 20 and at most 66 EVA letters with best-corrected vision, at each Screening visit.
7. The participant's study eye must have a HVF 24-2 SITA Standard visual field using spot size III with mean deviation -5 dB or worse and with a visual field defect compatible with NAION in the study eye (criteria in the MOP).

Exclusion Criteria (Cohort A):

1. The participant has received treatment for cancer within 12 months prior to enrollment (excluding localized basal cell carcinoma or localized squamous cell carcinoma) or had past diagnosis of cancer adjacent to the afferent visual pathway or had past diagnosis of metastatic cancer.
2. The participant had surgery, requiring general anesthesia with intubation, within 30 days prior to enrollment.
3. The participant is pregnant or a woman of child-bearing potential not using an acceptable method of contraception (per Section 4.1 of the protocol).
4. The participant is breast-feeding or plans to breast-feed.
5. The participant has had treatment with drugs that have potential neuroprotective or toxic effects on the optic nerve or retina (e.g., ethambutol, amiodarone, linezolid, hydroxychloroquine, fingolimod, brimonidine) within 6 months prior to enrollment.
6. The participant has participated in another interventional clinical trial within 60 days prior to enrollment, or previously participated in another clinical trial of RPh201 at any time.
7. The participant has been receiving or has received within three months prior to enrollment, corticosteroids (except topical steroids, steroid inhalers or intermittent injections into a joint or back), or immunosuppressive drugs.
8. The participant has a medical condition, social or psychological issue, or other condition which, in the judgment of the investigator, could be a safety concern or preclude the individual from completing the protocol.
9. The participant has a known allergy to cottonseed oil.
10. The participant is planning to move and not relocate near a study site and is unwilling to travel for appointments.
11. The participant cannot self-administer or arrange for administration of the IP.
12. The participant has one or more of the following abnormal test results at screening:

    * Erythrocyte Sedimentation Rate (ESR) above age/2 for men or [age + 10]/2 for women, as measured by Westergren method or equivalent.
    * Platelets >400,000 mm3
    * C-reactive protein (CRP) greater than two times the laboratory upper limit of normal.
    * Severe anemia (Hgb < 10)
13. The participant has symptoms, signs, and/or diagnosis of giant cell arteritis at any time.
14. The participant has any other optic neuropathies (e.g., optic neuritis or glaucoma) in either or both eyes (other than self-limited optic neuropathies in the non-study eye, such as past traumatic optic neuropathy or past transient steroid-induced glaucoma due to localized steroid administration).
15. The participant has systemic inflammatory or infectious disease associated with optic neuropathy or ocular disease.
16. The participant has a history of uveitis in the study eye within the last 10 years.
17. The participant's study eye has an ocular condition that appears consistent with a reduction in visual acuity to <20/25, diabetic retinopathy beyond mild non-proliferative diabetic retinopathy not involving the macula, or vision-threatening macula disease.
18. The participant has a visual field defect with homonymous non-altitudinal features or a defect that respects the vertical meridian.

Inclusion Criteria (Cohort B):

1. The participant must be 50 years of age or older at the time of the NAION episode in the study eye. This means that the participant's age at enrollment must be greater than or equal to the sum of 50 plus the number of years since NAION (e.g., at least 52 years of age if the episode was two years prior).
2. The participant must understand the nature of the procedure and provide written informed consent prior to any study procedure.
3. The participant has a definitive clinical diagnosis of NAION in the study eye that developed at least 6 months and no more than 3 years before randomization. Specifically, the disc swelling must have been observed and documented (by examination, OCT or photograph) by an ophthalmologist or neuro-ophthalmologist who previously examined the participant at the time of the NAION episode in the study eye during the acute episode.
4. The participant's study eye must have disc pallor (global or segmental) present.
5. The participant's study eye must have stable visual acuity (see Sections 5.3.3 and 5.3.4).
6. Using the study eye, the participant must read at least 20 and at most 66 EVA letters with best-corrected vision, at each Screening visit.

Exclusion Criteria (Cohort B):

1. The participant has received treatment for cancer within 12 months prior to enrollment (excluding localized basal cell carcinoma or localized squamous cell carcinoma) or had past diagnosis of cancer adjacent to the afferent visual pathway or had past diagnosis of metastatic cancer.
2. The participant had surgery, requiring general anesthesia with intubation, within 30 days prior to enrollment.
3. The participant is pregnant or a woman of child-bearing potential not using an acceptable method of contraception (per Section 4.1 of the protocol).
4. The participant is breast-feeding or plans to breast-feed.
5. The participant has had treatment with drugs that have potential neuroprotective or toxic effects on the optic nerve or retina (e.g., ethambutol, amiodarone, linezolid, hydroxychloroquine, fingolimod, brimonidine) within 6 months prior to enrollment.
6. The participant has participated in another interventional clinical trial within 60 days prior to enrollment, or previously participated in another clinical trial of RPh201 at any time. Participants who were randomized into the placebo arm of Cohort A of this protocol are eligible for screening for Cohort B.
7. The participant has been receiving or has received within three months prior to enrollment, corticosteroids (except topical steroids, steroid inhalers or intermittent injections into a joint or back), or immunosuppressive drugs.
8. The participant has a medical condition, social or psychological issue, or other condition which, in the judgment of the investigator, could be a safety concern or preclude the individual from completing the protocol.
9. The participant has a known allergy to cottonseed oil.
10. The participant is planning to move and not relocate near a study site and is unwilling to travel for appointments.
11. The participant cannot self-administer or arrange for administration of the IP.
12. The participant has one or more of the following abnormal test results at screening:

    1. Erythrocyte Sedimentation Rate (ESR) above age/2 for men or [age + 10]/2 for women, as measured by Westergren method or equivalent.
    2. Platelets >400,000 mm3
    3. C-reactive protein (CRP) greater than two times the laboratory upper limit of normal.
    4. Severe anemia (Hgb < 10 g/dL)
13. The participant has symptoms, signs, and/or diagnosis of giant cell arteritis at any time.
14. The participant has any other optic neuropathies (e.g., optic neuritis or glaucoma) in either or both eyes (other than self-limited optic neuropathies in the non-study eye, such as past traumatic optic neuropathy or past transient steroid-induced glaucoma due to localized steroid administration).
15. The participant has systemic inflammatory or infectious disease associated with optic neuropathy or ocular disease.
16. The participant has a history of uveitis in the study eye within the last 10 years.
17. The participant's study eye has an ocular condition that appears consistent with a reduction in visual acuity to <20/25, diabetic retinopathy beyond mild non-proliferative diabetic retinopathy not involving the macula, or vision-threatening macula disease.
18. The participant has a visual field defect with homonymous non-altitudinal features or a defect that respects the vertical meridian.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2020-09-27 (Actual); Study Completion 2020-09-27 (Actual)

PRIMARY OUTCOMES:
The change in number of best-corrected visual acuity (BCVA) letters from baseline to Week 26 (Cohort A) measured using electronic visual acuity (EVA). | Week 26 or Week 12
  Visual acuity
The change in number of best-corrected visual acuity (BCVA) letters from baseline to Week 12 (Cohort B) measured using electronic visual acuity (EVA). | Week 12
  Visual acuity

SECONDARY OUTCOMES:
The proportion of study eyes improving by a 15-letter score or more in BCVA from baseline to Week 26 using EVA (Cohort A). | Week 26
  Visual acuity
The proportion of study eyes improving by a 15-letter score or more in BCVA from baseline to Week 12 (Cohort B). | Week 12
  Visual acuity
The proportion of study eyes improving from baseline in five or more locations of the Humphrey visual field (HVF) 24-2 full-threshold with the size V stimulus on the glaucoma change probability map (GCPM) at the 5% level by group. | Week 26
  Humphrey visual field (HVF)
The proportion of study eyes improving by a 10-letter score or more in BCVA from baseline to Week 26 (Cohort A) using EVA. | Week 26
  Visual acuity
The proportion of study eyes improving by a 10-letter score or more in BCVA from baseline to Week 12 (Cohort B) using EVA. | Week 12
  Visual acuity

OTHER OUTCOMES:
The change in sensitivity on HVF-24-2 full-threshold with the size V stimulus. | Week 26
  Humphrey visual field (HVF)
The change in number of BCVA letters | Week 52
  Visual acuity
The proportion of study eyes improving by a 10-letter score or more in BCVA from baseline using EVA. | Week 52
  Visual acuity
The proportion of study eyes improving by a 15-letter score or more from baseline in BCVA by group. | Week 52
  Visual acuity
The mean change in sensitivity from baseline on HVF 24-2 full-threshold with the size V stimulus. | Week 52
  Humphrey visual field (HVF)
The proportion of study eyes improving in five or more locations from baseline of the HVF 24-2 full-threshold with the size V stimulus by GCPM at the 5% level by group. | Week 52
  Humphrey visual field (HVF)
The proportion of study eyes improving in mean deviation by 7 dB or more measured with HVF 24-2 SITA using the size III stimulus. | Week 12
  Humphrey visual field (HVF)
The proportion of study eyes improving by 7 dB or more in five or more locations measured with HVF 24-2 SITA using the size III stimulus. | Week 12
  Humphrey visual field (HVF)
The change in mean deviation measured with HVF 24-2 SITA using the size III stimulus. | Week 12
  Humphrey visual field (HVF)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard A Levin, M.D., Ph.D., Study Chair — McGill University
Locations (15):
- United States (15):
  - Byers Eye Institute at Stanford University, Palo Alto, California
  - UCLA Doheny Eye Center, Pasadena, California
  - The Eye Care Group, Orange, Connecticut
  - The Eye Care Group, Waterbury, Connecticut
  - Anne Bates Leach Eye Hospital/Bascom Palmer Eye Institute, Miami, Florida
  - Emory University, Atlanta, Georgia
  - NorthShore Medical Group, Glenview, Illinois
  - Bethesda Neurology, LLC, Rockville, Maryland
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Washington University Ophthalmology, St Louis, Missouri
  - New York Eye and Ear Infirmary of Mount Sinai, New York, New York
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Charleston Neuroscience Institute, Ladson, South Carolina
  - Neuro-Eye Clinical Trials, Inc., Houston, Texas
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available.

REFERENCES:
- [Background] Rath EZ, Hazan Z, Adamsky K, Solomon A, Segal ZI, Levin LA. Randomized Controlled Phase 2a Study of RPh201 in Previous Nonarteritic Anterior Ischemic Optic Neuropathy. J Neuroophthalmol. 2019 Sep;39(3):291-298. doi: 10.1097/WNO.0000000000000786. PMID 31430268
- See also: Randomized Controlled Phase 2a Study of RPh201 in Previous Nonarteritic Anterior Ischemic Optic Neuropathy — https://insights.ovid.com/crossref?an=00041327-201909000-00001